CLINICAL TRIAL: NCT00170521
Title: The Molecular Epidemiology of Streptococcus Pyogenes Among Children in Leon, Nicaragua
Brief Title: Mol Epi GrAS in Nicaragua
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0018; Leon GrAS2000
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2006-12

CONDITIONS: Streptococcus Group A
Keywords: group A streptococci, pharyngitis, epidemiology, Streptococcus pyogenes, children, Nicaragua
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine the epidemiology of throat isolates of group A streptococci among 3-15 year-old children with pharyngitis (sore throat) living in Leon, Nicaragua.

DETAILED DESCRIPTION:
Streptococcus pyogenes (GrAS) is a human pathogen that leads to great disease burden throughout the world. In the United States, an estimated 30 million infections occur yearly. Most of these are local infections of the skin or the throat but still lead to considerable use of health-care resources. These common, simple forms of GrAS disease may progress to or be followed by the more serious GrAS-related illnesses acute rheumatic fever, post-streptococcal glomerulonephritis, streptococcal toxic shock syndrome, sepsis, pneumonia, or other invasive illnesses. Outside the U.S., in the developing world, the burden of GrAS-related disease is presumed to be even higher, but is not completely elucidated in many of the poorer regions of the world. It is known, though, that rheumatic heart disease causes more cardiovascular morbidity in the children of the world than any other illness. Although the incidence of rheumatic fever in the U.S. has fallen to levels of approximately 0.5 per 100,000 per year, in some areas, the developing world's children still have rates over 100 per 100,000 per year. The percentage of cardiac admissions attributable to rheumatic heart disease in hospitals located in the developing world remains in the range of 30 to 50%, where it has been studied. GrAS is one of the best characterized human pathogens with regards to its microbiology, its spectrum of diseases, and its ability to lead to serious sequelae such as rheumatic fever and glomerulonephritis. Yet, efforts to control it through the use of antibiotics have been only partially successful in the United States and largely unsuccessful in the developing world. The health impact of uncomplicated streptococcal infections, such as pharyngitis, and the less common but more severe diseases, such as rheumatic heart disease, must be better studied in order to move forward with control measures. In this study, patients aged 3-15 presenting with sore throat, fever and cervical lymphadenopathy will be examined and a throat swab will be submitted to the lab for culture. All of these patients will be treated with either benzathine penicillin or, if they have a history of allergy to penicillin, oral erythromycin. The parent will be given a follow-up appointment to convey the result of the culture and to evaluate the course of the child's illness. Children presenting with sore throat only will be cultured and given a follow-up appointment to return after the result of the culture is known. Antibiotic treatment is given only if the culture is positive for group A streptococci. Within this algorithm is latitude for the physician to treat any patient based on clinical signs and symptoms and the concern that a particular child may not return for treatment if it is delayed based on the culture result. The overriding goal is the prevention of acute rheumatic fever and suppurative complications. The primary objective of this study is to characterize the GrAS isolates genotypically (emm type or sub-type). The secondary objective is to describe the epidemiology of throat isolates of GrAS among 3- to 15- year old children with pharyngitis living in Leon, Nicaragua. Primary endpoint of the study is the frequency and proportion of each emm-type among children with pharyngitis. Secondary Endpoints for the study are as follows: The proportion of children with pharyngitis from whom GrAS is isolated. The minimal incidence of GrAS pharyngitis in children based on annual cases per 100,000 children in the catchment areas. The age, gender, and ethnicity-specific minimal incidence rates of GrAS pharyngitis in children living in the catchment areas.

ELIGIBILITY:
Inclusion Criteria:

1. All children 3- to 15-years old with pharyngitis who are seen at a participating site will be invited to participate.

Exclusion Criteria:

1. Subjects whose parents are unable or unwilling to provide informed consent will be excluded from the study.
2. Children who are 13 years or older and unable or unwilling to provide informed consent will be excluded form the study.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13000
Dates: Start 2006-08; Study Completion 2008-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Autonomous University of Nicaragua, Leon, León, Nicaragua